CLINICAL TRIAL: NCT00288015
Title: An Open Label Multicenter Phase II Study of Bevacizumab for the Treatment of Angiosarcoma
Brief Title: Bevacizumab in Treating Patients With Angiosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Agulnik, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04S1; NU 04S1 (Other: Northwestern University); STU00006784 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma | interventions — Bevacizumab; Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab treatment until disease progression or intolerance
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab 15 mg/kg IV infusion given on day 1 every 21 days = (1 cycle).
  Other Names: rhuMAb; VEGF; Avastin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well bevacizumab works in treating patients with angiosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the median progression-free survival, in terms of stable disease, of patients with newly diagnosed or recurrent/refractory angiosarcoma treated with bevacizumab.

Secondary

* Evaluate the treatment effect of bevacizumab on the objective response rate as assessed by modified RECIST criteria in patients with angiosarcoma.
* Evaluate the duration of response.
* Assess the treatment effect of bevacizumab on duration of overall survival.
* Explore the objective response by target tumor density changes on CT scan.
* Evaluate the safety and tolerability of bevacizumab in patients with angiosarcoma.

OUTLINE: This is an open-label, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 to 4 months for 2 years.

PROJECTED ACCRUAL: A total of 31 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed angiosarcoma

  * Any stage disease
  * Must be deemed not surgically resectable (complete resection) and/or no other therapeutic modality is known to be curative
  * No angiosarcoma of a vessel wall
* Newly diagnosed or recurrent/refractory disease
* No prior tumor-related hemorrhage (any grade)
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* No CNS disease, brain metastases, or primary brain tumors

PATIENT CHARACTERISTICS:

* ECOG performance status of 0 or 1
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 gm/dL (transfusion and epoetin alfa allowed)
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Urine protein:creatinine ratio ≤ 1.0
* Total bilirubin ≤ 1.5 mg/dL
* Aspartate aminotransferase < 5 times ULN
* Alkaline phosphatase < 5 times ULN
* PT/INR ≤ 1.5 times ULN
* PTT ≤ 1.5 times ULN
* Fertile patients must use effective contraception
* Ejection fraction > 49% for patients with prior anthracycline therapy, ischemic cardiac disease, or history of heart failure
* No uncontrolled active infection
* No uncontrolled high blood pressure (defined as > 150/100 mm Hg)
* No symptomatic congestive heart failure (New York Heart Association class II-IV), unstable angina, cardiac arrhythmia, or myocardial infarction within the past 6 months
* No psychiatric illness or social situation that would limit study compliance
* No serious, nonhealing wound, ulcer, or bone fracture
* No evidence of bleeding diathesis or coagulopathy
* No clinically significant peripheral vascular disease
* Not pregnant or nursing
* No seizures not controlled with standard medical therapy
* No embolic or hemorrhagic stroke or prior transient ischemic attack
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No significant traumatic injury within the past 6 weeks

PRIOR CONCURRENT THERAPY:

* No prior therapy with bevacizumab or other antiangiogenesis treatment
* No major surgical procedure or open biopsy within the past 6 weeks
* No more than 2 prior chemotherapy regimens
* No fine-needle aspiration or core-needle biopsy or other minor surgical procedure within the past 7 days
* No radiotherapy within the past 28 days
* No concurrent chronic daily treatment with aspirin > 325 mg/day or nonsteroidal anti-inflammatory medications
* No concurrent warfarin or any other anticoagulant (any dose)
* No concurrent radiotherapy
* No concurrent major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-10; Primary Completion 2013-06-06 (Actual); Study Completion 2016-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agulnik, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on June 1, 2005 with an accrual goal of up to 31 patients. The study was designed to enroll 12 patients initially and do an interim efficacy assessment. Accrual was suspended on February 28, 2007 for this analysis and reopened on May 15, 2007. Study was closed to accrual permanently on April 19, 2010.
Period: Registered to Study
Arm/Group | Bevacizumab
Started | 32
Completed | 32
Not Completed | 0
Period: Bevacizumab Treatment Cycles 1-2
Arm/Group | Bevacizumab
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: First Response Assessment
Arm/Group | Bevacizumab
Started | 30
Completed | 26
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Physician Decision | 2
Period: Continued Bevacizumab Cycle 3+
Arm/Group | Bevacizumab
Started | 26
Completed | 19
Not Completed | 7
Not completed — Disease progressed | 7
Period: Follow up for Survival x 2 Years
Arm/Group | Bevacizumab
Started (Includes all patients who received bevacizumab cycle 1 and were still living.) | 29
Completed | 3
Not Completed | 26
Not completed — Death | 13
Not completed — Lost to Follow-up | 4
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
Type of Sarcoma [Count of Participants; unit: Participants]
  angiosarcoma | 24
  epitheliod hemangioendothelioma | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival of Patients Treated With the Study Drug as Defined by RECIST Criteria.
Description: During treatment, tumor assessment was done by MRI scan after the second cycle of study treatment, after the forth cycle of study treatment, and then every 3 cycles of treatment thereafter. After Study drug completion, tumor assessment by MRI was done every 3 to 4 months (for up to 2 years after the last bevacizumab dosage).
  Responses were categorized according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.0.
  Progressive Disease (PD) was defined as having at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: After cycles 2 and 4, then every 3 cycles thereafter while on treatment (1 cycle = 21 days); every 3-4 months after treatment up to 2 years.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Bevacizumab
Number analyzed (Participants) | 30
Weeks | 12.4 [10.1 to 14.76]
Statistical Analysis 1: Comparison: Bevacizumab; This is a two stage optimal simon design testing the Null hypothesis: bevacizumab is not effective with P<=0.220 and the alternative hypothesis: bevacizumab is effective with P >=0.450 and has a sample size of 16.96 and a probability of early termination of 0.739. p=probability (progression free survival - PFS time>/=3 months); Test type: Other — This is a two-stage optimal simon design. If bevacizumab is not effective, there is a 0.050 probability of concluding that it is. If bevacizumab is effective, there is a 0.2000 probability of concluding that it is not; Kaplan-Meier estimate — In first stage 12 patients will be entered, if </=3 patients have PFS time>3 months p</=0.22 is likely true. In second stage a total of up to 31 patients data will be analysed. If >/=10 patients show PFS</=3 months, it will suggest p>0.50 is true; P<=0.220 is the threshold value of significance that the null hypothesis is true or the alternative hypothesis is true. P Value was not calculated from the data. Median survival time was calculated using a 20% censored Kaplan-Meier table and graph

2. Secondary Outcome: Objective Response Rate in Patients Treated With Bevacizumab.
Description: Objective response rate will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  Stable Disease, neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
  Progressive Disease, defined as having at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 30
Participants
  Partial response | 4
  Stable disease | 15
  Progressive disease | 11

3. Secondary Outcome: Duration of Response.
Description: During treatment, evaluation of response will be done by MRI scan after the second cycle of study treatment, after the forth cycle of study treatment, and then every 3 cycles of treatment. After Study drug completion, evaluation of response will be assessed by MRI every 3 to 4 months (for 2 years after the last bevacizumab dosage).
Time Frame: as for outcome 1
Population: Data for this outcome measure was not collected. By the time the results of the study were being collected, this outcome measure was no longer relevant as Recist 1.0 was in use. As a result, data for this outcome measure was not collected or analysed. Time to progression was a more relevant data point.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess the Treatment Effect of Bevacizumab on Duration of Overall Survival
Description: After Study drug completion, assessment of treatment effect of bevacizumab on duration of overall survival will be assessed by MRI every 3 to 4 months (for 2 years after the last bevacizumab dosage).
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Bevacizumab
Number analyzed (Participants) | 30
Weeks | 107 [44.29 to 169.99]

5. Secondary Outcome: Evaluate the Toxicity of Bevacizumab.
Description: Toxicity data for bevacizumab will be collected on day 1 of every cycle (1 cycle = 21 days) during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Day 1 of every cycle, on average every 21 days until end of treatment up to 2 years.
Population: Number of participants with either grade 1 (mild), 2 (moderate),3 (severe), 4 (life-threatening) adverse event related to treatment.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 30
participants
  Participants with one bevacizumab related event | 26
  Thromboyctopenia | 4
  Shortness of breath | 5
  Hypertension | 7
  Pain | 3
  Nausea | 5
  Infection | 2
  Headache | 4
  Anemia | 6
  Decline in FEV1 | 1
  Hyperglycemia | 1
  Transient ischemic attack | 1
  Neuromotor function | 2
  Cardiac (congestive heart failure) | 1
  Plural effusion | 1
  Liver-clinical | 1
  Anorexia | 2
  Fatigue | 9
  Alopecia | 3
  Dizziness | 2
  Edema | 2
  Dementia | 1
  Hemorrhage (epitasis) | 1

6. Post Hoc Outcome: Time to Progression
Description: During treatment, tumor assessment was done by MRI scan after the second cycle of study treatment, after the forth cycle of study treatment , and then every 3 cycles of treatment thereafter. After Study drug completion, tumor assessment by MRI was done every 3 to 4 months (for up to 2 years after the last bevacizumab dosage) Responses were categorized according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.0.
  Progressive Disease (PD) was defined as having at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: After cycles 2 and 4, then every 3 cycles thereafter while on treatment (1 cycle = 21 days); ever 3-4 months after treatment up to 2 years
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Bevacizumab
Number analyzed (Participants) | 30
Weeks | 26 (53)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 5 year period.
Arm/Group | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 14/30
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=30)
Cardiac ( congestive heart failure) (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Bladder infection (urinary) (Infections and infestations) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) — resulting in a fall
Speech impairment (Nervous system disorders) | 1 (1) — Episode of inability to speak
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (non cardiac) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Knee surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Shot in leg (Social circumstances) | 1 (1) — Patient shot himself in the leg
Upper respiratory - bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=30)
Fatigue (General disorders) | 17 (23)
Headache (Nervous system disorders) | 10 (18)
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 9 (16)
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 5 (10)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Platelet decrease (Blood and lymphatic system disorders) | 7 (16)
hypertension (Cardiac disorders) | 15 (24)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia- atrial fibrillation (Cardiac disorders) | 2 (2)
Fever (General disorders) | 4 (4)
Insomnia (General disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Weight loss (General disorders) | 5 (7)
Partial Thromboplastin Time (PTT) (Investigations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Ascites (non malignant) (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (Gastrointestinal disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (17)
salivary gland changes (metallic taste) (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9)
difficulty swallowing (dysphagia) (Gastrointestinal disorders) | 1 (1)
Nose bleed (Hemorrhage) (General disorders) | 5 (7)
upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Colon infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Edema (limbs) (Blood and lymphatic system disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (12)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Chest pain (General disorders) | 1 (1)
High glucose (hyperglycemia) (Metabolism and nutrition disorders) | 4 (5)
low glucose (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
High potassium (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Sensory neuropathy (Nervous system disorders) | 6 (7)
Dizziness (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
CNS cerebrovascularischemia - Transient ischemic attack (Nervous system disorders) | 1 (1) — (Transient ischemic attack)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice change/alteration (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Blurred vision (Eye disorders) | 2 (2)
Watery eye (Eye disorders) | 1 (3)
Urine color change (Renal and urinary disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Flu-like syndrome (General disorders) | 3 (6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (General disorders) | 3 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
AST, SGPT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 7 (11)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 7 (8)
Decline in FEV1 (forced expiratory volume) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 2 (2) — Night sweats
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
anorexia (Gastrointestinal disorders) | 8 (9)
Alkaline phosphatase increase (Metabolism and nutrition disorders) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes